CLINICAL TRIAL: NCT06701825
Title: A Multicentre, Controlled, Randomised and Single-blind, Adaptive Phase IV Protocol to Evaluate Effectiveness and Cost-effectiveness of Pre-emptive Genotyping Strategy to Optimise Tacrolimus Dosage in a Pretransplant Chronic Kidney Disease Population Cohort
Brief Title: Effectiveness and Cost-effectiveness of a Pre-emptive Genotyping Strategy in Patients Receiving Tacrolimus
Acronym: TRANSPGx
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto de Investigación Hospital Universitario La Paz (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-516596-32-00; 2024-516596-32-00 (EU CTIS Number)
Record Dates: First submitted 2024-11-20; First posted 2024-11-22 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Kidney Disease, Chronic; Transplant Recipient (Kidney); Immunosuppression
Keywords: Tacrolimus; Kidney transplant; Cost-effectiveness; Pharmacogenetic; Phase IV Clinical Trial
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Tacrolimus

STUDY DESIGN:
Intervention Model Description: Phase IV, multicentre, controlled, randomized, parallel and single-blind adaptive clinical trial nested within the iPHARMGx master protocol study
Who Masked: Participant
Masking Description: Subjects will remain blinded to arm assigned because pharmacogenetic phenotype and tacrolimus dose-guidance will only be exclusively accesible to the attending physician
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of care (Active Comparator): Patients in this control group will receive treatment with any formulation of Tacrolimus authorized and commercialized in Spain. They will be administered tacrolimus according to clinical practice and the drug's product labeling.
  Interventions: Drug: Tacrolimus
- Dose adjusted by guidelines (Experimental): Participants in this experimental group will receive treatment with any formulation of Tacrolimus authorized and commercialized in Spain. They will be administered the specific dosage of tacrolimus recommended by the Clinical Pharmacogenetics Consortium's genotype guidelines, utilizing the patient's pharmacogenetic information and characteristics.
  Interventions: Drug: Tacrolimus

INTERVENTIONS:
Drug: Tacrolimus — Tacrolimus at the dosage reccomended by the "Clinical Pharmacogenetics Implementation Consortium (CPIC) Guidelines for CYP3A5 Genotype and Tacrolimus Dosing" based on the subjects pharmacogenetic phenotype.
  Arms: Standard of care
Drug: Tacrolimus — Subject allocated to this arm will receive tacrolimus according to clinical practice and the drug's product labelling. These subject will not receive a personalised dose based on their pharmacogenetic phenotype.
  Arms: Dose adjusted by guidelines

SUMMARY:
This is a phase IV multicentre adaptive single-blinded randomized clinical trial to evaluate if preemptively genotyping populations at pretransplant chronic kidney disease susceptible of receiving tacrolimus therapy is effective, cost-effective, and feasible within the Spanish National Health System when compared to the current standard of care. This trial is nested within the iPHARMGx master protocol.

DETAILED DESCRIPTION:
This is a nation-wide, multicentre, randomised, controlled, and adaptive phase IV clinical trial that aims to assess the effectiveness and cost-effective of pre-emptive pharmacogenetic testing strategies, including those impacted by genetic variants associated with adverse drug reactions (ADRs) or limited efficacy. The clinical trials will evaluate the effective and cost-effective of pre-emptive genotyping by defining a drug-gene-endpoint triad. Study subjects will be pre-emptively genotyped and, if found to have an actionable gene variant, randomly allocated to either a test group where guideline-based treatment modifications will be initiated or a control group that will be managed according to healthcare provider standard of care (SoC). Subsequently, subjects will be prospectively followed at prespecified timepoints. Detailed information on drug-gene-endpoint triads, allocation schemes, and follow-up visits will be provided in each of the subprotocols. A Data Monitoring Committee (DMC), composed of physician experts, will be appointed for each nested trial to review the data on an ongoing basis, ensuring the safety of participants and scientific validity of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be willing and able to provide written informed consent prior the initiation of any study procedures.
2. Subject or their legally authorized representative has voluntarily signed the informed consent document.
3. Participant is on the waiting list for a kidney transplant.
4. Subject is able and willing to take part and be followed-up for the majority of the study duration, and adhere to the procedures specified in this protocol.
5. Subjects must be naïve to any genotyping test of the following genes: CYP3A5.

Exclusion Criteria:

1. Known hypersensitivity/allergy reaction to tacrolimus or any of the excipients.
2. History of renal, heart, and/or liver transplant.
3. History or clinical evidence of any disease and/or existence of any surgical or medical condition, which might interfere in a relevant manner with the absorption, distribution, metabolism, or excretion of the study treatment, except for renal disease.
4. Any condition or situation precluding or interfering the compliance with the protocol.
5. Any condition at medical discretion for which renal transplantation and/or study treatment should not be received.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2025-06-02 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Tacrolimus concentrations levels | 4 days
  Number and percentage of patients achieving tacrolimus target plasma concentrations at visit 3. Tacrolimus concentrations levels at day 4 (+/-1d) will be the effectiveness surrogate outcome. It will be considered therapeutic range levels between 7-10 ng/ml.

SECONDARY OUTCOMES:
Incremental cost-effectiveness ratio (ICER) | Though study completion, on average 18 months
  Cost-effectiveness ratio that divides the differences in costs between both treatments by the difference in effectiveness between both treatments.
Number and percentage of patients with transplant rejection. | Though study completion, on average 18 months
  Transplant rejection will be considered if there is histological confirmation and/or the patient initiates any type of therapy aimed at treating rejection (e.g. corticosteroids).
Rate of AE associated to treatment. | Though study completion, on average 18 months
  All adverse events associated to tacrolimus will be recorded during the study
Number and percentage of patients achieving tacrolimus target plasma concentrations at visit 4, 5 and 6. | Week 4, 15 and 26
Healthcare expenditure related to predefined events of interest | Though study completion, on average 18 months
  Any costs made as a result of an AE
Incidence of discontinuation or treatment modification | Though study completion, on average 18 months
  Incidence of discontinuation or treatment modification due to lack of effective related to the drug of inclusion.

OTHER OUTCOMES:
Novel prognostic and predictive genetic biomarkers of tacrolimus safety and effectiveness | Though study completion, on average 18 months
  All participants DNA sample will be susceptible of deep sequencing analysis assessed trough techniques only available at Nation Centre of Oncological Investigations (CNIO) and genome-wide association studies when applicable
Identification of new actionable genes/relevant polymorphisms within the predefined population subsets | Though study completion, on average 18 months

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital La Paz, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
A copy of the database of data collected during the clinical trial will be attached as an appendix to the publication resulting from this clinical trial.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available at the same time as the results will be published, and will be kept available to everyone without any time limit.
Access Criteria: Data will be available indefinitely on the publisher's website, as long as it is kept by the Publisher, for anyone who wishes to access the data, for non-commercial purposes.